CLINICAL TRIAL: NCT04678986
Title: Emergency Room Evaluation for Older Users of Emergency Departments: Predicting Adverse Health Outcomes With Deep Learning Algorithms
Brief Title: ER2 and Deep Learning for Prediction of Adverse Health Outcomes
Status: Withdrawn | Type: Observational
Why Stopped: Study not begun in time and has been withdrawn because of feasibility
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Olivier Beauchet, Professor of Geriatrics, Jewish General Hospital
Other Study IDs: 2021-2699
Record Dates: First submitted 2020-12-14; First posted 2020-12-22 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Emergencies
Keywords: Geriatrics; Emergency rooms; adverse health events prevention; Deep learning
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ER2 participants: all participants of ER2 database will be included in the analysis
  Interventions: Other: ER2

INTERVENTIONS:
Other: ER2 — No intervention, data analysis only

SUMMARY:
An Emergency Department (ED) visit for an older adult is a high-risk medical intervention. Known adverse events (AE) include delirium, prolonged ED or hospital stay, hospitalization, recurrent ED visits and hospital death. These happen in a growing proportion in ED visitors over age 65 are over who are represented in ED visits.

Tools predicting AEs in the ED are of paramount importance to help decision-making on patient triage and disposition. They can help identify areas of unmet needs for seniors in order to develop targeted actions. Multiple scoring systems including "Programme de recherche sur l'intégration des services de maintien de l'autonomie" (PRISMA-7), Identification of Seniors at Risk (ISAR), Clinical Frailty Scale (CFS), Brief Geriatric Assessment (BGA) have extensively been studied in the ED and other settings for various outcomes. These tools rely on a simple scoring system that minimally trained staff can reliably and quickly administer. Doing otherwise is unlikely to be applicable to daily clinical practice.

As prediction accuracy has not significantly improved in the past decade, perhaps new analysis strategies are necessary. The current hype surrounding deep learning comes from better and cheaper hardware and the availability of simple and open-source libraries supported by large companies and a broad community of users. Hence, implementing deep learning (DL) algorithms is now open to a wide range of settings, including medical care in a standard clinical practice. DL has been shown to be more accurate than the average board-certified specialist on very specific tasks. Prediction of various clinical outcomes has produced less dramatic results, perhaps as traditional (non-DL) models already outperformed clinicians for many disease states. Published DL approaches applied to outcome prediction in the ED have focused on acutely ill adults in general, specific conditions or administrative issues such as admitting department or ED overcrowding. None have targeted a specific age group like older ED visitors.

An important caveat to many DL approaches is interpretation of results. To develop interventions based on targeted features associated with AEs in a given model, it has to be somewhat transparent. If multiple layers of NNs improve prediction compared to linear regression, they often provide no clinically relevant insight on how and which variables interact to yield that result.

ELIGIBILITY:
Inclusion Criteria:

* Age above 75 years old
* Unplanned Emergency department visit

Exclusion Criteria:

* Do not meet inclusion criteria

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Between September 2017 and July 2020, 47 000 Emergency Department visits met the selection criteria. Training DL models on tabular data has been shown to be less effective than on unstructured sources such as images or sound. An appropriate mitigation strategy is to increase the quantity of data. Hence, all participants of the ER2 database will be included in the analysis. All visits will be included in the analysis.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-02-24 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
ED length of stay | through database constitution, from September 2017 to July 2020
  The length of emergencey department stay is defined as the average number of hours that patients spend in Emergency department.

SECONDARY OUTCOMES:
Prolonged hospital stay | through database constitution, from September 2017 to July 2020
  The prolonged length of hospital stay is defined as a stay above the average number of days that patients spend in hospital
Number of partciipants with at least one hospitalizations | through database constitution, from September 2017 to July 2020
  Defined as the admission in hospital after an admission in Emergency department
recurrent ED visits | through database constitution, from September 2017 to July 2020
  Defined as all the Emergency department recurrent visit within 30 days
Number of partciipants with diagnosis of delirium | through database constitution, from September 2017 to July 2020
  Defined as a diagnosis of delirium in teh medical chart of the patient
Number of partciipants with hospital death | through database constitution, from September 2017 to July 2020
  Defined as a reported death during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Beauchet, MD, Principal Investigator — McGill University
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No